CLINICAL TRIAL: NCT01956383
Title: Phase III of Study of Safety and Efficacy of the PrePex Device for MC Programs in Zimbabwe (Nurses Study)
Brief Title: Safety and Efficacy of the PrePex Device Circumcision When Performed by Nurses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ministry of Health and Child Welfare, Zimbabwe (Other)
Responsible Party: Principal Investigator, Prof. Mufuta Tshimanga, Public Health Physician, Department of Community Medicine, University of Zimbabwe, Ministry of Health and Child Welfare, Zimbabwe
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MRCZ/A/1628 Nurses Study
Record Dates: First submitted 2012-09-19; First posted 2013-10-08 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Circumcision Adult; HIV CDC Category B2
Keywords: male circumcision; HIV; Zimbabwe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PrePex™ device (Experimental): Adult male circumcision by the PrePex™ device
  Interventions: Device: PrePex™ device

INTERVENTIONS:
Device: PrePex™ device — PrePex™ device for adult male circumcision. The PrePex™ device facilitates adult male circumcision that is bloodless with no anesthesia and no sutures

SUMMARY:
The protocol, approved by the Medical Research Council, was issued to assess the safety and efficacy of the non-surgical device for applying it to the national scale up of adult male circumcision in Zimbabwe

DETAILED DESCRIPTION:
Models show that to have the highest impact on the HIV epidemic, circumcision of up to 80% of men in high prevalence countries, where MC rates are low, needs to be achieved (UNAIDS 2009; Manicaland HIV/STD Prevention Project, 2008; Bollinger, et al, 2009). Hallett and colleagues in 2008 showed that for Zimbabwe specifically, HIV incidence could be reduced between 25% to 35% if about 50% of men are circumcised. All modelings conducted show that MC programs must be part of a comprehensive HIV prevention package as MC alone will not tip the HIV epidemic into a terminal decline.

The PrePex Device offers hope for rapid scale up of adult male circumcision in resource limited settings.

Once the safety and efficacy have been established, it is important to conduct operations research to determine how best to implement both device and surgical circumcisions in the national program. Thus, the Zimbabwe MOHCW is planning a three phase trial in order to determine the safety of the PrePexTM device, its performance and the ease of use in an implementation roll out.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 30 years
* Uncircumcised
* Wants to be circumcised
* Agrees to be circumcised by any of the study methods ,PrePex or Surgical as appropriate
* HIV sero-negative
* Able to understand the study procedures and requirements
* Agrees to abstain from sexual intercourse and to keep caution not to directly rub the cut area if masturbating, for 8 weeks post removal (9 weeks total)
* Agrees to return to the health care facility for follow-up visits (or as instructed) after his circumcision for a period of 8 weeks post removal (9 weeks total)
* Subject able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have good compliance for the study
* Subject agrees to anonymous video and photographs of the procedure and follow up visits
* Agrees to stay overnight at the Hospital in order to follow pain measurements in the first 16 hours

Exclusion Criteria:

* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the subject from undergoing a circumcision
* HIV sero-positive
* Subject with the following diseases/conditions: phimosis, paraphimosis, warts under the prepuce, torn or tight frenulum, narrow prepuce, hypospadias, epispadias
* Known bleeding / coagulation abnormality
* Uncontrolled diabetes
* Subject that to the opinion of the investigator is not a good candidate
* Subject does not agree to anonymous video and photographs of the procedure and follow up visits
* Refusal to take HIV test.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 603 (Actual)
Dates: Start 2012-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To assess the safety of the PrePex device when circumcision is performed by nurses | 9 weeks
  To assess the safety of the PrePex device by means of the following parameters: Clinical significant adverse event rate when circumcision is performed by nurses

SECONDARY OUTCOMES:
Evaluate the training needs of PrePexTM deployment using nurses | 9 weeks
  1. PrePex Procedure time and the resulting cost of provider's time
  2. Cost Effectiveness • Cost of device
  3. Evaluation of the PrePex training needs and efficacy
  4. Acceptability of the PrePex procedure by the patients
Observation of in-field usability of device | 9 weeks
  Observation of in-field usability of device using questionnaires
Obtain user feedback from nurses | 9 weeks
  Obtain user feedback from nurses by questionnaires
Assess safety compared to physician deployment | 9 weeks
  1. To assess the safety of the PrePex device by means of the following parameters: Clinical significant adverse event rate, when circumcision is performed by nurses comparing to Physicians.
Assess practicality and acceptability among nurses and patients | 9 weeks
  Assess practicality and acceptability among nurses and patients using questionnaires.
Assess satisfaction of procedure among nurses and patients | 9 weeks
  Assess satisfaction of procedure among nurses and patients using questionnaires.
Determine cost-effectiveness compared to surgical procedure | 9 weeks
  1. Evaluating the cost-effectiveness when taking into account the following parameters: i. PrePex Procedure time and the resulting cost of provider's time compared to surgical procedure ii. Cost of device compared to surgical procedure iii. Cost of device training compared to surgical procedure training iv. Cost of staff time for follow-up visits compared to compared to surgical procedure staff time v. Cost of equipment and supplies needed for the circumcision procedure for both PrePex and surgical circumcision.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Gwinji, MBChB, MPH, Principal Investigator — PS- MoHCW
Locations (1):
- Znfpc Spilhaus Center, Harare, Zimbabwe

REFERENCES:
- See also: MRCZ — http://www.mrcz.org.zw/